CLINICAL TRIAL: NCT03877302
Title: The Effect of Reflexology on Labor: A Randomized Controlled Experimental Study
Brief Title: The Effect of Reflexology on Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Semra Çevik, phD, Assiatant Professor, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017/159
Record Dates: First submitted 2019-03-04; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Reflexology
Keywords: Birth; Reflexology; Pain
MeSH Terms: conditions — Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: A total of 60 women participated in the study in 2 groups of 30 for reflexology and control groups. By giving appropriate position in the first stage of delivery to the pregnant women in the experimental group, 10-minute massage was applied to both feet including 5-minute massage for each foot starting first from the right foot by using vaseline under the supervision of a doctor to facilitate the hand movements, then the reflexology technique was applied by stimulating the nerve points by applying pressure to reflex regions of each foot for 20 minutes as totally 40 minutes for both feet. The control group was composed of pregnant women who received routine treatment, care and applications of the hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reflexology group (Experimental): In addition to providing routine nursing/midwifery care, foot reflexology was applied by the researcher to the pregnant women in the experimental group in the active phase of labor (dilatation 4 cm). By giving appropriate position to the pregnant women, the massage was done to both feet for totally 10 minutes including 5 minutes for each foot starting from right foot under the supervision of a doctor. Whereupon, the reflexology technique was applied by stimulating the nerve points by applying pressure to reflex regions of each foot for 20 minutes as totally 40 minutes for both feet. As reflex points of the feet for manual pressure in labor pain; 1: Solar Plexus, 2: Hypothalamus, 3: Pituitary, 4: Spleen, 5: Thyroid Gland, 6: Adrenal, 7: Intestine, 8: Spinal Cord 9: Uterus, Vagina, Ovaries and Fallopian Tubes were studied.
  Interventions: Other: reflexology
- Control Group (No Intervention): The control group received only routine treatment, care, and practices of the hospital. Visual Analog Scale (VAS) and State-Trait Anxiety Inventory (STAI FORM TX-I) were evaluated 2 times as in active (4-7 cm) and transition (8-10 cm) phases in the pregnant women in the control group. After the delivery, the Birth Satisfaction Scale was applied to the women by the researcher.

INTERVENTIONS:
Other: reflexology — foot reflexology
  Arms: reflexology group

SUMMARY:
Aims and Objectives: The purpose of this study was to determine the effect of reflexology, one of the non-pharmacological methods used in the management of labor pain, on anxiety, labor duration, labor pain, and labor satisfaction in primiparous pregnant women.

Background: Labor pain is one of the most severe types of pain experienced by a woman throughout her life. As a result of the labor pain and birth-related stress, maternal and fetus health is negatively affected. Controlling of labor pain will decrease the anxiety and tension experienced by pregnant woman.

Design: A randomized controlled experimental was used. Method: A total of 60 women participated in the study in 2 groups of 30 for reflexology and control groups. By giving appropriate position in the first stage of delivery to the pregnant women in the experimental group, 10-minute massage was applied to both feet including 5-minute massage for each foot starting first from the right foot by using vaseline under the supervision of a doctor to facilitate the hand movements, then the reflexology technique was applied by stimulating the nerve points by applying pressure to reflex regions of each foot for 20 minutes as totally 40 minutes for both feet. The control group was composed of pregnant women who received routine treatment, care and applications of the hospital.

DETAILED DESCRIPTION:
Aims:This study was conducted as a randomized controlled experimental study in order to determine the effect of reflexology application in primiparous pregnant women on labor pain, anxiety, labor duration, and birth satisfaction.

METHOD Participants The study was conducted with voluntary pregnant women applying to the delivery room unit of Gaziantep Cengiz Gökçek Maternity and Children Hospital to perform their first birth between 01 July 2017 and 07 July 2018. When the sample volume that would represent the population with the conditions of α= 0.05 risk, 1-α =0.95 accuracy rate, B= 0.20, 1-B= 0.80 power ratio was considered with the comparison results of VAS mean scores in the study by Dolation et al., it was determined to be minimum 27 people for each group.

The study was conducted with two groups including Reflexology Group (experimental) and Control Group. By including 30 women into each group, the study was conducted with a total of 60 women. The drawing method was used to decide to which group the women would be assigned. In order to draw lots, 60 small paper pieces were prepared, control was written on 30 of these paper pieces, reflexology was written on the other 30 pieces of paper, and they were then folded and placed into a bag. Inclusion of women into groups was determined according to the papers women drew from the bag.

Data Collection Tools The data of the study were collected using "Descriptive Information Form", "Visual Analog Scale (VAS)", "State-Trait Anxiety Scale (STAI FORM TX-I )", and "Birth Satisfaction Scale".

Descriptive Information Form: The form prepared by the researcher by examining the related literature consists of two sections. In the first section, age, height, weight, educational level, and working status of the woman along with the number of birth, parity, number of abortus, number of living children, and modes of previous births were asked. The second section of the form includes questions related to the period of birth stages (Stages I, II, and III), interventions made in the first stage of birth and during the labor (Oxytocin administration, amniotomy, Fundal pressure, Vacuum etc.), perineal tear, Apgar score and the newborn's status of being accepted to the intensive care unit.

Visual Analog Scale (VAS): Visual Analogue Scale (VAS) is used to describe the severity of pain in patients with pain. The diagnosis will be established based on subjective data including the patient's verbal expression. There are numbers horizontally placed varying from 0 to 10. The pain severity is expressed in numbers ranging from 0 to 10 and no pain is determined with "0" and the most severe pain is determined with "10". In this method, it is explained that there are two endpoints and she is free to mark any point between these two points.

State-Trait Anxiety Inventory: To determine state and trait anxiety levels of the participants, the state-trait anxiety inventory (STAI FORM TX -I) was used. The individual is required to indicate the feelings or behaviours that he/she has experienced in a specific situation according to the degree of severity by marking one of the options such as (1) Never, (2) Little, (3) Very and (4) Completely. The state-trait anxiety inventory requires the individual to describe how he/she feels at a certain moment and under certain conditions by considering his/ her feelings about a specific situation. While high scores indicate high anxiety levels, low scores indicate low anxiety levels. The state-trait anxiety inventory consists of 20 statements. The score obtained from the scale may vary between 20 and 80. While a high score represents a high anxiety level, a low score represents a low anxiety level.

Birth Satisfaction Scale: Birth Satisfaction Scale was developed by Martin and Fleming in 2009. The original language of the scale is English. The translation of the scale was performed by Coşar et al.,. The scale is a Likert-type scale that is scored according to the responses. The scale form consists of 30 items and total score obtained from the scale varies between 30 and 150. As the scores obtained from the scale increase, birth satisfaction level increases.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who were 19 years old and older,
* Pregnant women who had singleton pregnancy, were between 38-42nd weeks of gestation,
* Pregnant women who can perform spontaneous vaginal delivery,
* Pregnant women who were at the beginning of the active phase in the first phase of action (4 cm dilatation),
* Pregnant women who were primiparous, can establish verbal communication,
* Pregnant women who agreed to participate in the study.

Exclusion Criteria:

* Pregnant women who had risky pregnancy,
* Pregnant women who had a systemic disease that would interfere with normal birth,
* Pregnant women who were in the second stage of labor

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 60 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-07 (Actual); Study Completion 2018-07-07 (Actual)

PRIMARY OUTCOMES:
VAS scores | 6 hours
  Visual Analogue Scale (VAS) was used to measure the severity of labour pain. The diagnosis will be established based on subjective data including the patient's verbal expression. There are numbers horizontally placed varying from 0 to 10. The pain severity is expressed in numbers ranging from 0 to 10 and no pain is determined with "0" and the most severe pain is determined with "10". In this method, it is explained that there are two endpoints and she is free to mark any point between these two points Analog Scale (VAS) was evaluated 2 times as active (4-7 cm) and transition (8-10 cm) phases after reflexology application.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory | 6 hours
  The State Anxiety Inventory requires the individual to describe how she feels at a certain moment and under certain conditions by considering her emotions about the situation she is in. While high scores refer to high anxiety levels, low scores indicate low anxiety levels. The state anxiety inventory consists of 20 expressions. The score value obtained from the scale varies between 20 and 80 points. While high score indicates high anxiety level, low score shows low anxiety level. In scoring made according to the criteria directive, 0-19 points are evaluated as "none", 20-39 points as "mild", 40-59 points as "moderate", 60-79 points as "severe", and 80 points as "severe anxiety".The State -Trait Anxiety Inventory (STAI FORM TX-I) was evaluated 2 times as active (4-7 cm) and transition (8-10 cm) phases after reflexology application.

OTHER OUTCOMES:
Birth Satisfaction | 1 hour
  The scale form consists of 30 items and total score obtained from the scale varies between 30 and 150. As the scores obtained from the scale increase, birth satisfaction level increases.Birth Satisfaction Scale was applied by the researcher to the women after the delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Semra Çevik, phD, Principal Investigator — University of Gaziantep
Locations (1):
- Gaziantep University, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No